CLINICAL TRIAL: NCT04902703
Title: Phase II Trial to Evaluate Safety and Efficacy of GM-CSF/Sargramostim in Alzheimer's Disease (SESAD)
Brief Title: Phase II Trial to Evaluate Safety and Efficacy of GM-CSF/Sargramostim in Alzheimer's Disease
Acronym: SESAD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Alzheimer's Association (Other); Partner Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-2727; 1R01AG071151-01 (NIH)
Record Dates: First submitted 2021-05-14; First posted 2021-05-26 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer; Alzheimers Disease; sargramostim; GM-CSF; Leukine
MeSH Terms: conditions — Alzheimer Disease | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Water

STUDY DESIGN:
Intervention Model Description: The study is double-blind, placebo-controlled in the Alzheimer's Disease population, and will include individuals with mild AD and moderate AD. Individuals who meet inclusion/exclusion criteria will be randomized in a double-blind manner, to receive either sargramostim 178. 57µg/m2/day subcutaneously (7 days per week) or placebo (7 days per week) in an approximate 2:1 randomization ratio.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sargramostim (Experimental): 178.57 mcg/m2/day subcutaneously 7 days/week for 24 weeks
  Interventions: Drug: Sargramostim
- Placebo Control - Saline (Placebo Comparator): Placebo comparator (saline) subcutaneously 5days/week for 24 weeks
  Interventions: Drug: Saline - placebo comparator

INTERVENTIONS:
Drug: Sargramostim — Sargramostim is a granulocyte macrophage colony stimulating factor that will be administered at a dose of 178.57 mcg/m2 per day subcutaneously, 7 days/week, for 24 weeks
  Other Names: Leukine; Granulocyte Macrophage Colony Stimulating Factor
  Arms: Sargramostim
Drug: Saline - placebo comparator — Saline will be administered subcutaneously, 7 days/week, for 24 weeks
  Other Names: Sterile solution of sodium chloride in water
  Arms: Placebo Control - Saline

SUMMARY:
A medicine that is FDA-approved for bone marrow stimulation (called sargramostim) will be tested for its safety and efficacy in individuals with mild-to-moderate Alzheimer's disease over a six month treatment period.

DETAILED DESCRIPTION:
This trial protocol is designed to evaluate primarily whether the long-term use of sargramostim (recombinant human GM-CSF), administered five days per week for six consecutive months (24 weeks), will be tolerated by and safe for use in participants with mild-to-moderate AD, secondarily whether sargramostim can slow, halt, or reverse cognitive decline, and exploratory whether sargramostim can slow, halt, or reverse decline in activities of daily living, reverse or improve several biomarkers associated with AD, as evaluated by multimodal neuroimaging techniques and blood and cerebrospinal fluid analyses. This trial extends the safety results from recently completed Phase 2 double-blind, placebo-controlled clinical trial in mild-to-moderate AD participants (NCT01409915, COMIRB#12-1273), using sargramostim that was administered five days per week for three consecutive weeks and in which there were no incidence of drug-related serious adverse events (SAEs).

ELIGIBILITY:
Inclusion Criteria:

* Males or females between age 60 and 85 years, inclusive, at time of consent.
* Have a dedicated partner/caregiver informant who is in the company of the participant at least 12 hours a week, who can accompany them to scheduled visits, and who is able to provide accurate reporting upon the behavioral, cognitive and functional abilities of the participant.
* Be physically able to participate with adequate visual acuity and auditory discrimination.
* Be willing / able to provide written informed consent or assent.
* Must reside within a proximity of the study site that will not preclude their regularly-scheduled participation in the trial, as well as a catchment area for local lab blood draws (i.e. central contracted laboratory).
* Meet criteria for probable AD dementia according to the National Institute of Aging - Alzheimer's Association (NIA-AA) 2018 core research criteria, and have the following at screening:

  * A diagnosis of mild AD or moderate AD, or
  * A provisional research diagnosis consistent with probable mild AD or moderate AD, and
  * MoCA score of 4-24 inclusive.
* Have positive biomarker for brain amyloid pathology as shown by:

  * Positive plasma assay for Aβ(42)/ Aβ(40) ratio AND
  * Either postivie CSF assay for AD assessment or positive amyloid PET, per PI read.
* If receiving anti-dementia treatment (i.e. AChEI), be on stable treatment for at least 2 months (i.e., cholinesterase inhibitor and/or Memantine) before initial screening visit.
* Be stable on all other medications for at least 30 days prior to initial screening visit.

Exclusion Criteria:

* Individuals with a first degree relative diagnosed with AD before 55 years of age.
* BMI ≥35.
* Is unable to read/write at an appropriate level to reliably participate in clinical trial psychometric assessments.
* Is a prisoner.
* Other neurological or psychiatric condition (other than AD) that can impact cognition, as well as atypical presentations of AD and AD related dementias, including logopenic primary progressive aphasia (PPA), or posterior cortical atrophy (PCA); or, CT/MRI evidence of potentially significant intracranial abnormalities not related to AD (e.g., evidence of major stroke or lacune in an area critical to cognition, infections, cancer, hydrocephalus, multiple sclerosis, etc.); or abnormal CSF not consistent with AD.
* Presence of current, serious mood or anxiety disorder, and/or a psychotic disorder, and/or a substance-related disorder according to Diagnostic and Statistical Manual of Psychiatric Disorders, Edition IV, text revision (DSM-IV-TR) or DSM-V that, in the opinion of the Principal Investigator, might impact cognitive assessment, affect participants ability to complete the study, or confound interpretation of the study drug effect; or is considered suicidal or shows suicidal ideation as assessed by the study physician
* History of deep vein thrombosis, pulmonary embolism, familial predisposition for deep vein thrombosis, or pulmonary embolism.
* Active cancer / malignant neoplasm within 5 years of screening other than non-melanoma skin cancers (e.g. Basal cell or squamous cell). Previous diagnosis of Leukemia, despite remission state or length of time, is considered exclusionary.
* History of a latex or yeast allergy.
* Presence/history of drug hypersensitivity; or known hypersensitivity to sargramostim, yeast-derived products, any other component of the product, or benzyl alcohol (present in bacteriostatic water or saline for injection).
* History of asplenia, hyposplenia, or splenectomy
* History of, or treatment for, an autoimmune disease (e.g. Rheumatoid Arthritis, Multiple Sclerosis, Myasthenia Gravis, etc.).
* Untreated or unstable medical condition that could interfere with the study assessments in the opinion of the study physician, or may require immune-stimulating, immune-suppressive, or immune-modulating treatment(s) during the conduct of the study.
* History of seizures (except infant febrile seizures).
* Pregnant or breastfeeding female, or female of childbearing potential and not protected by highly effective contraceptive method of birth control (i.e., oral or depot contraceptives or intrauterine device (IUD) or participant was surgically sterilized) and/or unwilling or unable to be tested for pregnancy; Male refusing to use condoms, if partner can get pregnant.
* MRI evidence of >4 micro-hemorrhages; participants who may be prone to spontaneous ARIA-H and/or may be more susceptible to adverse effects of the ARIA-H.
* Laboratory results that are, in the judgement of the investigator, indicative of an untreated medical or hematologic condition that could increase risk or interfere with study assessments
* Evidence of:

  * Clinically significant pre-existing fluid retention (clinical or radiological);
  * respiratory symptoms (e.g., dyspnea), moderate-to-severe lung disease (e.g. COPD, pulmonary infiltrates)
  * cardiovascular symptoms or electrocardiographic evidence of cardiac disease that warrant therapeutic intervention (e.g., congestive heart failure, supraventricular arrhythmia, heart block, uncontrolled atrial fibrillation, etc.)
  * a resting pulse less than 50, as reviewed by the study physician;
  * prolonged QTc interval >470 ms in females, 450 ms in males).
  * screening blood pressure measurement of greater than 160 systolic and/or 95 diastolic
* Known renal dysfunction or serum creatinine >150 μmol/L, or Glomerular Filtration Rate (GFR) less than 55 ml/min
* Known hepatic dysfunction (apart from Gilbert's syndrome) or serum ALT ≥3 times the upper limit of normal (ULN)
* Positive serology for hepatitis B surface antigen (HBs Ag), anti-hepatitis C virus (anti-HCV), anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti-HIV2 Ab) or spirochetal infection (e.g. syphilis)
* Contraindication to lumbar dural puncture, including coagulopathy, concomitant anticoagulation therapy (except daily 81 mg aspirin), prior spinal surgery, significant deformity of the lumbar/sacral region, or any other factor that, in the opinion of the investigator, precludes safe LP procedure.
* Contraindication or inability to complete magnetic resonance imaging (e.g., cardiac pacemaker/defibrillator, ferromagnetic metal implants) or PET scan.
* Sensitivity to fluorodeoxyglucose F 18
* Having past or planned exposure to ionizing radiation that would, together with the radiation resulting from the administrations of the PET tracer(s) used in this study, exceed applicable institutional, local, or national recommendations for annual or lifetime exposure.
* Poor venous access.
* Chronic use of no-n-steroidal anti-inflammatory drugs (NSAIDs), excepting 81 mg daily aspirin therapy or acetaminophen.
* Taking any prohibited medication or therapy
* Be the recipient of an investigational drug within 60 days of screening, or within 5 times the elimination half-life of that drug, whichever is the longest.
* Prior treatment with an investigational anti-amyloid or anti-tauopathy therapy, or AD vaccine, unless it can be documented that they were on placebo.
* Participation in the treatment phase of an investigational sargramostim clinical trial within 6-months of screening.
* Any interested participant who:

  1. Is in the judgement of the Principal Investigator likely to be non-compliant with study protocol, including, but not limited to, leaving the area of the study for any extended period; or separate from the designated caregiver/informant, without acceptable replacement, for any of the scheduled assessment visits during the study.
  2. Is unable to cooperate because of a language problem or because of a developmental disability.
  3. Oversees or implements any aspect of the study, or is employed by Partner Therapeutics or its affiliates or subsidiaries, or is an employee of the University of Colorado Alzheimer's and Cognition Center and is engaged in the conduct of the study, or first degree relative of such.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by number of Adverse Events (AEs) by body system | Informed consent to Follow-up Visit (38 weeks)
  The safety of sargramostim will be assessed through number of adverse events (AEs) by body system from consent to follow-up within a safety analysis set consisting of all individuals who were enrolled and and randomized and who received at least on injection of sargramostim or placebo.

SECONDARY OUTCOMES:
Mini-Mental State Examination | Baseline to End of Treatment, Follow-up (30 weeks)
  Mini-Mental State Examination (MMSE) is a brief psychometric instrument developed to assess cognitive function in elderly populations. It is a standard assessment used by all NIH Alzheimer's Disease Centers (ADCCs and ADRCs) to identify and monitor individuals with AD. The range for scores in the MMSE is from 0 to 30, with lower scores indicating greater impairment.

OTHER OUTCOMES:
Alzheimer's Disease Assessment Scale - cognitive subscale (ADAS-Cog13) | Baseline to End of Treatment, Follow-up (30 weeks)
  The ADAS-Cog13 measures the severity of the most important symptoms of AD. and consists of 13 tasks measuring the disturbances of memory, language, praxis, attention and other cognitive abilities. , which are often referred to as the core symptoms of AD. The score ranges form 0-85, with higher score denoting worse performance
Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB) | Baseline to End of Treatment, Follow-up (30 weeks)
  The CDR is a study partner/caregiver and participant based interview to assess changes in domains such as memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Each domain is rated as 0 (no dementia), 0.5 (uncertain dementia), 1 (mild dementia), 2 (moderate dementia), or 3 (severe dementia). Range is 0-18. Higher scores denote worse functioning
Trail Making Test - Part A (TMT-A) | Baseline to End of Treatment, Follow-up (30 weeks)
  Psychomotor speed will be assessed by the Trail Making Test-A, a timed test in which participants must connect a series of numbers randomly placed on a page. Time range is 0-150 seconds, with a higher time denoting worse performance
Alzheimer's Disease Cooperative Study -Activities of Daily Living Inventory (ADCS-ADL) | Baseline to End of Treatment, Follow-up (30 weeks)
  The ADCS-ADL is a caregiver/study partner rated questionnaire of 23 items, with possible scores over a range of 0-78, where 78 implies full functioning with no impairment.
Montreal Cognitive Assessment (MoCA) | Baseline to End of Treatment, Follow-up (30 weeks)
  The Montreal Cognitive Assessment (MoCA) is a brief, assessment developed for detection and tracking of cognitive impairment and is sensitive for detecting Alzheimer's disease. Measuring multiple domains, it is commonly used in both clinical and research settings, and is well validated, with a range of scores from 0-30.
Neuropsychiatric Inventory (NPI) | Baseline to End of Treatment, Follow-up (30 weeks)
  Neuropsychiatric Inventory (NPI) is a study partner/caregiver interview to assess any changes in neuropsychiatric status in such domains as hallucinations, delusions, agitation, depression, anxiety, disinhibition, apathy and aberrant motor behaviors. It assesses presence of symptoms, and scores by severity X frequency (Range 0-12 in each symptom category), and caregiver distress (Range 0-5). The higher the scores, the the greater the presence of the impact of the symptom.
Verbal Fluency | Baseline to End of Treatment, Follow-up (30 weeks)
  Verbal fluency (producing words that start with a specific letter of the alphabet, also known as letter fluency) is a timed test where a participant produces as many works as they can in 60 seconds. The more correct words that a participant produces, the higher the score.
Semantic Fluency | Baseline to End of Treatment, Follow-up (30 weeks)
  Semantic fluency (producing words that belong in a category, such as animals, also known as category fluency) is a timed test where a participant produces as many works as they can in 60 seconds within a category. The more correct words that a participant produces, the higher the score.
Exploratory: Fluorodeoxyglucose Positron Emission Tomography (FDG PET) assessment of brain metabolism | Baseline to End of Treatment (24 weeks)
  FDG-PET assessment of metabolic activity, overall, as well in different brain regions, particularly in the medial temporal lobe in potential correlation with changes in MTA

CONTACTS AND LOCATIONS:
Overall Officials: Huntington Potter, PhD, Principal Investigator — University of Colorado Alzheimer's and Cognition Center
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Potter H, Woodcock JH, Boyd TD, Coughlan CM, O'Shaughnessy JR, Borges MT, Thaker AA, Raj BA, Adamszuk K, Scott D, Adame V, Anton P, Chial HJ, Gray H, Daniels J, Stocker ME, Sillau SH. Safety and efficacy of sargramostim (GM-CSF) in the treatment of Alzheimer's disease. Alzheimers Dement (N Y). 2021 Mar 24;7(1):e12158. doi: 10.1002/trc2.12158. eCollection 2021. PMID 33778150
- See also: CU Alzheimer's and Cognition Center Clinical Research Portal — http://www.cumemoryresearch.org

DOCUMENTS (5):
  • Study Protocol (2025-07-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT04902703/Prot_000.pdf
  • Informed Consent Form: Optional PET (2025-06-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT04902703/ICF_001.pdf
  • Informed Consent Form: Optional LP (2025-06-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT04902703/ICF_002.pdf
  • Informed Consent Form: Participant (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT04902703/ICF_003.pdf
  • Informed Consent Form: study partner ICF (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT04902703/ICF_004.pdf